CLINICAL TRIAL: NCT07244328
Title: An Exploratory Clinical Trial of UX-GIP001 Injection (Human GABAergic Interneuron Progenitor Cells Injection) in Adult Patients With Drug-Resistant Unilateral Mesial Temporal Lobe Epilepsy
Brief Title: Exploratory Study of UX-GIP001 Cell Therapy in Adult Patients With Drug-Resistant Unilateral Mesial Temporal Lobe Epilepsy (MTLE)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shanghai UniXell Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0876
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy; MTLE
Keywords: Unilateral Medial Temporal Lobe Epilepsy (MTLE); GABAergic Inhibitory Interneuron Progenitor Cells; Drug-Resistant Epilepsy (DRE)
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: open-label, single-center, dose-escalation and dose-expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UX-GIP001 (Experimental): Two dose levels will be planned. Each patient only receives one corresponding dose of UX-GIP001.
  Interventions: Biological: UX-GIP001

INTERVENTIONS:
Biological: UX-GIP001 — Allogeneic human GABAergic interneuron precursors (UX-GIP001) are delivered into the temporal lobe region of the brain.

SUMMARY:
This is an exploratory clinical trial (Protocol: UX-GIP001-101) investigating UX-GIP001 Injection, a novel cell therapy product consisting of human GABAergic interneuron progenitor cells (GIP), for treating adult patients with drug-resistant unilateral medial temporal lobe epilepsy (MTLE). The primary objective is to assess the safety, tolerability, and preliminary efficacy of UX-GIP001. This is an open-label, single-arm study. All enrolled participants will receive the active investigational cell therapy. Seizure frequency and safety parameters will be evaluated by comparing post-transplant outcomes to pre-transplant baselines.

DETAILED DESCRIPTION:
Participants will receive UX-GIP001 via stereotactic neurosurgery, preceded by and followed with immunosuppressive therapy. The study includes a baseline period for eligibility confirmation and a 24-month follow-up phase involving regular safety assessments, neuroimaging , seizure diary logging, and evaluations of quality of life, cognition, and mood. This pioneering regenerative approach seeks to provide a new treatment strategy for drug-resistant MTLE by addressing the underlying pathophysiology.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 18-75 (inclusive), male or female.
2. Clinical presentation consistent with unilateral mesial temporal lobe epilepsy (MTLE).
3. Has failed to achieve seizure control despite treatment with at least two anti-seizure medications (ASMs) at recommended or maximally tolerated doses.
4. Average focal seizure frequency ≥4 per 28 days during the 3 months prior to screening.
5. Stable doses of ASMs for ≥1 month prior to enrollment.
6. Patient is in good general health or has stable comorbid conditions, and has adequate organ function.

Key Exclusion Criteria:

1. Epilepsy caused by other/or progressive neurological diseases , or patients experiencing only focal aware seizures without observable manifestations.
2. History of epilepsy surgery.
3. History of status epilepticus within 12 months prior to screening.
4. Presence of long-term implants in the skull or intracranial space.
5. Severe systemic disease or dysfunction.
6. Primary or secondary immunodeficiency.
7. History of clear suicidal intent, plan, or behavior within one year prior to screening.
8. Severe psychiatric disorders.
9. History of malignancy within the past 5 years, except for cervical carcinoma in situ, basal cell or squamous cell skin cancer cured for >5 years.
10. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs)/Serious Adverse Events (SAEs) | From baseline to 2 years post surgery

SECONDARY OUTCOMES:
Change from baseline in total and subtype seizure frequency | From baseline to 2 years post surgery
Responder rates (≥50% and ≥75% reduction) in total and subtype seizure frequency | From baseline to 2 years post surgery
Seizure free rate | From baseline to 2 years post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Wang, Doctor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Junming Zhu, Doctor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No